CLINICAL TRIAL: NCT02858596
Title: The Effect of Semi-solid Feeding After Percutaneous Endoscopic Gastrostomy (PEG) on Clinical Outcomes, Specifically the Incidence of Aspiration Pneumonia and Postoperative Length of Stay
Brief Title: The Effect of Semi-solid Feeding After Percutaneous Endoscopic Gastrostomy (PEG) on the Incidence of Aspiration Pneumonia and Postoperative Length of Stay
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hiroshima Kyoritsu Hospital (Other)
Responsible Party: Principal Investigator, Wong Toh Yoon, Chief Gastroenterologist, Hiroshima Kyoritsu Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Semi-solid trial
Record Dates: First submitted 2016-08-01; First posted 2016-08-08 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Gastrostomy; Aspiration Pneumonia
MeSH Terms: conditions — Pneumonia, Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Semi-solid feed group (Experimental): Given semi-solid feed protocol
  Interventions: Dietary Supplement: Semi-solid feed (Terumo PG soft)
- Liquid feed group (Placebo Comparator): Given liquid feed protocol
  Interventions: Dietary Supplement: Liquid feed (Meibalance)

INTERVENTIONS:
Dietary Supplement: Semi-solid feed (Terumo PG soft)
  Arms: Semi-solid feed group
Dietary Supplement: Liquid feed (Meibalance)
  Arms: Liquid feed group

SUMMARY:
Percutaneous endoscopic gastrostomy (PEG) is a minimally invasive procedure for long-term enteral tube feeding in patients with insufficient oral intake. Although peristomal site infection is often noted as the most common adverse event after PEG tube placements, it is seldom life-threatening and considered a minor adverse event. Feeding-related adverse events have been identified as the main cause of death after PEG, with up to 50% of postoperative early mortality (30 days) being attributed to aspiration pneumonia. This may be related to the persistence of gastroesophageal reflux (GER) of enteral feed after gastrostomy, even though PEG have been demonstrated to be superior to nasogastric tube feeding in terms of preventing GER. It has been more than a decade since semi-solid feeds were developed as an alternative to conventional liquid feeds to prevent feeding-related adverse events. Unfortunately, there is limited published literature on this topic despite the wide usage of this feeding method in Japan. Amidst the growing popularity of this method and the introduction of National Healthcare Insurance coverage for semi-solid feed prescriptions, we initiated a semi-solid feed protocol along with our existing post-PEG feeding protocols in 2014.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving gastrostomy tube placement in our hospital for enteral nutrition.

Exclusion Criteria:

* Patients receiving gastrostomy tube placement for decompression
* Patients with no gut usage more than 2 weeks before procedure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Incidence of aspiration pneumonia | through study completion, average 90 days postoperation

SECONDARY OUTCOMES:
Postoperative length of stay | through study completion, average 90 days postoperation

CONTACTS AND LOCATIONS:
Overall Officials: Toh Yoon Wong, MD, Principal Investigator — Hiroshima Kyoritsu Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shizuku T, Adachi K, Furuta K, Niigaki M, Miyaoka Y, Katoh S, Kobayashi K, Otani M, Kawashima K, Otani J, Kinoshita Y. Efficacy of half-solid nutrient for the elderly patients with percutaneous endoscopic gastrostomy. J Clin Biochem Nutr. 2011 May;48(3):226-9. doi: 10.3164/jcbn.10-108. Epub 2011 Apr 13. PMID 21562643
- [Background] Adachi K, Furuta K, Morita T, Nakata S, Ohara S, Tanimura T, Koshino K, Miki M, Ishimura N, Inoue Y, Ryuko K, Umegae N, Ohhata S, Katoh S, Yamamoto K, Nariai Y, Hashimoto Y, Sumi A, Kawaguchi M, Kinoshita Y. Half-solidification of nutrient does not decrease gastro-esophageal reflux events in patients fed via percutaneous endoscopic gastrostomy. Clin Nutr. 2009 Dec;28(6):648-51. doi: 10.1016/j.clnu.2009.05.006. Epub 2009 Jun 5. PMID 19501431
- [Background] Nishiwaki S, Araki H, Shirakami Y, Kawaguchi J, Kawade N, Iwashita M, Tagami A, Hatakeyama H, Hayashi T, Maeda T, Saitoh K. Inhibition of gastroesophageal reflux by semi-solid nutrients in patients with percutaneous endoscopic gastrostomy. JPEN J Parenter Enteral Nutr. 2009 Sep-Oct;33(5):513-9. doi: 10.1177/0148607108327045. Epub 2009 Jun 1. PMID 19487579
- [Background] Tanishima Y, Fujita T, Suzuki Y, Kawasaki N, Nakayoshi T, Tsuiboi K, Omura N, Kashiwagi H, Yanaga K. Effects of half-solid nutrients on gastroesophageal reflux in beagle dogs with or without cardioplasty and intrathoracic cardiopexy. J Surg Res. 2010 Jun 15;161(2):272-7. doi: 10.1016/j.jss.2009.03.025. Epub 2009 Apr 19. PMID 19577758